CLINICAL TRIAL: NCT02319616
Title: A Randomized Placebo Controlled Split-body Double-blind Phase II Clinical Trial to Investigate the Safety and Efficacy of Clobetasol 0.05% Ointment for the Treatment of Toxic Epidermal Necrolysis (TEN)
Brief Title: Topical Clobetasol for the Treatment of Toxic Epidermal Necrolysis
Acronym: TEN
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804284
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Toxic Epidermal Necrolysis
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Clobetasol; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clobetasol 0.05% ointment (Experimental): All patients will have one arm assigned to receive the experimental treatment (topical clobetasol 0.05% ointment) applied daily for a period of fourteen days.
  Interventions: Drug: Clobetasol 0.05% ointment
- Placebo (Placebo Comparator): All patients will have one arm assigned to receive the placebo treatment (topical petrolatum ointment) applied daily for a period of fourteen days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clobetasol 0.05% ointment — Blinded, daily application to one arm for a period of fourteen (14) days
  Arms: Clobetasol 0.05% ointment
Drug: Placebo — Blinded, daily application to one arm for a period of fourteen (14) days
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to investigate the efficacy and safety of topical steroid ointment (clobetasol 0.05%) for the treatment of the cutaneous manifestations of toxic epidermal necrolysis (TEN).

DETAILED DESCRIPTION:
The experimental focus of this trial is thus to evaluate the safety and clinical outcomes of topical steroid (clobetasol 0.05% ointment) for treatment of the cutaneous manifestations of toxic epidermal necrolysis (TEN).

The design of the study is a randomized, placebo-controlled, double-blind split-body Phase II clinical trial in which clobetasol 0.05% or placebo ointment will be topically applied to opposite arms for a period of fourteen days. The primary endpoints of the study are to determine the time to cessation of skin detachment in both groups as well as the safety of topical clobetasol to treat the cutaneous manifestations of TEN. Secondary outcome measures will evaluate efficacy by comparing the time to re-epithelialization and the percentage of affected skin between the clobetasol and placebo arms at various time points.

An additional aim of the study is to characterize the genes expressed during the TEN disease state and any changes in gene expression following treatment with topical steroids, particularly those genes involved in the regulation of programmed cell death (apoptosis). This will be accomplished though molecular analysis of skin biopsy specimens obtained after treatment with clobetasol and placebo ointments. The specific hypothesis being tested is that two weeks of topical clobetasol will promote epidermal keratinocyte survival through suppression of TNF signaling, decreased granulysin expression and inhibition of other pro-apoptotic pathways resulting in shorter disease duration and decreased time to re-epithelialization.

IRB number: 642415-5

ELIGIBILITY:
Inclusion Criteria:

* Characteristic histological findings on diagnostic biopsy
* Clinical diagnosis verified by two independent physicians
* Greater than 10% affected body surface area (BSA)
* Ability to start treatment within seven days or less from the onset of erosions
* Actively worsening disease (enlarging area of involvement or new erosions occurring over the last 24 hours)
* Patient Body Surface Area (BSA) > 1.0 m2
* Reproductive age female patients must have a negative pregnancy test prior to enrollment

Exclusion Criteria:

* Patients will be excluded if they are < 7 or > 85 years of age.
* Patients who have documented:

  * Uncontrolled infection (e.g. documented bacteremia)
  * Malignancy
  * Known prior immunodeficiency
  * Pregnancy
  * Concurrent use of systemic corticosteroids in the burn center greater than or equal to 0.5 mg/kg/day of prednisone or equivalent dose of similar medication.
  * Greater than 70% eroded skin
  * SCORETEN score >3 on hospital admission
* Patients will also be excluded if they have: active hepatitis and/or an ALT or AST greater than four times the normal limits, or renal insufficiency with an estimated GFR<50 mL/min/1.73m2.

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Safety (numeric cellulitis score) | 14 days
  Local infection (cellulitis) is a potential complication of treatment with topical steroid ointment. A primary outcome measure of the study will be to determine if any difference in local infection rate exists between between control and clobetasol-treated skin in patients with toxic epidermal necrolysis, determined by daily assessments and assignment of a numeric cellulitis score.
Time to Cessation of Skin Detachment | 14 days
  The time until cessation of skin detachment (measured in days) will be determined though daily skin examinations and compared between the clobetasol and placebo-treated skin of patients with toxic epidermal necrolysis.

SECONDARY OUTCOMES:
Time to 90% re-epithelialization | 14 days
  The time to 90% re-epithelialization will be determined by daily skin examinations and recorded in days to determine if a significant difference exists between control and clobetasol treated skin.
Percent Affected Surface Area | 14 days
  Percent affected surface area will be measured with daily skin examinations and compared between the placebo and steroid treated skin in patients with TEN
Percent Affected Surface Area Detached Skin | 14 days
  The percent body surface area affected by detached skin will be monitored through daily skin examinations and compared between the clobetasol and placebo treated skin in patients with toxic epidermal necrolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilken R, Li CS, Sharon VR, Kim K, Patel FB, Patel F, Maverakis E. Topical clobetasol for the treatment of toxic epidermal necrolysis: study protocol for a randomized controlled trial. Trials. 2015 Aug 22;16:374. doi: 10.1186/s13063-015-0879-7. PMID 26297574